CLINICAL TRIAL: NCT07187245
Title: Reality PAWS: Examining the Feasibility of a Mixed Reality Dog Visitation Program for Hospitalized Children in Isolation
Brief Title: Feasibility of the Reality PAWS Program for Children in Isolation
Status: Not yet recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Children's Hospital Colorado (Other)
Collaborators: Children's Hospital Los Angeles (Other)
Responsible Party: Principal Investigator, Jennifer Staab, MS, CCLS, Principal Investigator, Children's Hospital Colorado
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Supportive Care
Other Study IDs: 25-1732
Record Dates: First submitted 2025-09-10; First posted 2025-09-22 (Actual); Last update posted 2025-09-22 (Actual); Status verified 2025-09

CONDITIONS: Inpatient Pediatric Care; Isolation; Feasibility Studies

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: Yes | US Export: No

ARMS (1):
- Reality PAWS VR Program Session on Meta Quest 3 VR Device (Experimental): Participants will be able to wear a Meta Quest 3 VR Device and interact with the Reality PAWS VR program for up to 30 minutes per session.
  Interventions: Device: Reality PAWS Program via Meta Quest 3 VR

INTERVENTIONS:
Device: Reality PAWS Program via Meta Quest 3 VR — Reality PAWS is a mixed reality (MR) game that allows patients to interact with a virtual dog. It was developed at Children's Hospital Colorado to serve patients under isolation precautions who are unable to be visited by a facility dog in person. Patients can interact with the game through features such as walking the dog, providing commands, outfitting the dog, giving treats, playing fetch, petting the dog, and playing with others.

SUMMARY:
The goal of this clinical trial is to learn if a mixed reality program, Reality PAWS, delivered on a Meta Quest 3 VR headset, is a feasible intervention for pediatric patients in isolation. It will also evaluate the safety of the program and its effect on pain, anxiety, and loneliness. The main questions the study aims to answer are:

What is the feasibility of utilizing Reality PAWS MR as a substitute for in-person dog therapy for children under isolation precautions? Are patients compliant with using Reality PAWS MR? What are the interventional outcomes of Reality PAWS MR?

Participants will:

Wear a Meta Quest 3 VR headset with the Reality PAWS program. Interact with the program. Answer surveys regarding demographics, anxiety, pain, loneliness, sickness, perceived exertion, and immersion in the program.

ELIGIBILITY:
Inclusion Criteria:

* Children 8 to 21 years old admitted to Children's Hospital Colorado or Children's Hospital Los Angeles
* Children who are English-speaking (legal guardian may be English-speaking or Spanish-speaking)
* Children within the normal range of development will be recruited for this study.

Exclusion Criteria:

* Traumatic brain injury, neurological disorders, neurodevelopmental issues, or other neurological disorders and comorbidities that may confound study outcomes and administration of the study protocol and metrics (e.g., visual field disturbances, frequent nausea/ vomiting, not medically stable, intellectual disability)
* Children with visual, auditory, or tactile deficits that would interfere with the ability to complete the experimental tasks
* Children with a history of seizure disorder
* Children currently sick with flu-like symptoms or experiencing a headache or earache
* Children with known or suspected motion sickness
* Children with cochlear implants or pace makers

Ages: 8 Years to 21 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult
Enrollment: 50 (Estimated)
Dates: Start 2025-10 (Estimated); Primary Completion 2026-04 (Estimated); Study Completion 2026-04 (Estimated)

PRIMARY OUTCOMES:
Recruitment Feasibility | Through study completion, an average of 6 months.
  Number of screened patients, number of eligible patients, number of enrolled patients, number of withdrawn patients, number of subsequent Reality Paws sessions received/requested by patients.
Intervention Feasibility - Time Spent Using MR | From baseline until study session completion, approximately 30 minutes.
  Time spent using MR.
Intervention Feasibility - Software | From baseline until study session completion, approximately 30 minutes.
  Number of technology or software issues.
Electonic Case Report Qualitative Feedback and Observations | From baseline until study session completion, approximately 30 minutes.
  Qualitative self-reported and observed experience on the electronic case report form related to patient's engagement in the MR.
Measurement Feasibility | Through study completion, an average of six months.
  Percent of participants who completed all surveys. This will be determined by taking the number of survey's completed and dividing it by the total number of survey's.
Child Simulator Sickness Questionnaire | Completed at baseline and again at study session completion, approximately 30 minutes after completing the study intervention MR.
  Assesses potential side effects of using Reality PAWS, children will provide ratings of simulator sickness using the 7-item Child Simulator Sickness Questionnaire. Consists of items related to potential side effects common to individuals after playing in virtual environments, such as "sickness, headache, and dizziness. The questionnaire asks about symptoms currently experienced as rated on a 0 - 2 scale, with 0 = No, 1 = A little, and 3 = A lot. There are three scoring categories: nausea, oculomotor, and disorientation, with specific questions falling under each category. Each category adds scores of three questions, and a score of three or more indicates simulator sickness.
Borg Rating of Perceived Exertion | At intervention session completion, approximately 30 minutes after starting the MR intervention.
  Children will rate their physical exertion after playing Reality PAWS using the Borg Rating of Perceived Exertion. This one-item scale consists of a single question asking children to rate their subjective feeling of exertion, without considering the kinds of physical demands that might lead to this feeling. The scale ranges from 6 (no exertion at all) to 20 (maximal exertion), with higher scores indicating higher levels of perceived exertion.
Gold-Rizzo Immersion and Presence | Completed at study session completion, approximately 30 minutes after completing the MR intervention.
  The Gold-Rizzo Immersion and Presence assesses three domains: sense of involvement, perceived realism, and sense of transportation within the software. The measure contains 16 questions where patients can respond either "no," "a little," or "a lot." Higher total scores indicate a higher level of immersion.
Amount of adverse or serious adverse events | Until study completion, about 6 months.
  Number of adverse and/or serious adverse events.

SECONDARY OUTCOMES:
Faces Anxiety Scale | Collected at baseline, before the intervention, and again after intervention, on average, 30 minutes after.
  Children will be asked to report their anxiety using the Faces Anxiety Scale before and after the MR session. The Faces Anxiety Scale is a single item scale with five possible responses ranging from a neutral face to one showing extreme fear.
Faces Pain Scale | Collected at baseline, before the intervention, and again after intervention, on average, 30 minutes after.
  The Faces Pain Scale - Revised (FPS-R) is a valid and reliable self-report measure where patients see a scale of 6 different faces representing various intensities of pain, ranging from "no pain" to "very much pain."
Childhood Anxiety Sensitivity Index | Collected at baseline, before the intervention, and again after intervention, on average, 30 minutes after.
  A modified version of the Anxiety Sensitivity Index, and is a self-report questionnaire which measures a child's belief that their anxiety will have negative consequences.
Loneliness Visual Analog Scale | Collected at baseline, before the intervention, and again after intervention, on average, 30 minutes after.
  Used to assess loneliness in children via a one-item, self-report, visual analog scale thermometer that includes faces as anchors. The question asks how lonely the child is feeling in the moment, on a rating scale from 0 being not lonely at all, and 10 being extremely lonely.
Multidimensional State Boredom Scale - Short Form | Collected at baseline, before the intervention, and again after intervention, on average, 30 minutes after.
  An eight question scale that is used for brief assessments of boredom. Participants are asked to rank their agreement with the statements using a 7-point Likert scale, 1= Strongly disagree, and 7= Strongly agree, with higher scores indicate higher levels of state boredom.

CONTACTS AND LOCATIONS:
Locations (2):
- United States (2):
  - Children's Hospital Los Angeles, Los Angeles, California
  - Children's Hospital Colorado Anschutz Medical Campus, Aurora, Colorado

IPD SHARING:
Plan to Share IPD: No